CLINICAL TRIAL: NCT00449397
Title: A Naturalistic, Prospective, Single Centre, Double Blinded, Fixed Dose, Randomised, Four Week Comparison Study Investigating Efficacy, Tolerability and Safety of 200 mg Per Day Versus 400 mg Per Day Quetiapine Fumarate in 200 Drug naïve First Episode Psychosis Patients Aged 15 to 25 Years.
Brief Title: Dose Finding of Quetiapine Fumarate 200mg vs 400mg in First Episode Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AU-SEA-0003
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Psychosis
Keywords: First Episode Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine Fumarate

SUMMARY:
The purpose of this study is determine the minimal effective dose and the impact on:

1. treatment outcomes at 4, 12 and/or 48 weeks the treatment has required to treat patients experiencing the first psychotic episode
2. the final maintenance doses
3. the use of other medications
4. the amount of changes to other antipsychotic medication
5. the number of hospitalization days

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing their first psychotic episode
* Male or Female
* Aged 15-25

Exclusion Criteria:

* Previous treatment with antipsychotic medication (longer than 1 week)
* History of a clinically significant physical illness
* Organic disorder presenting with psychotic symptoms

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Medication dose, Remission and response rate, exBPRSvs4, SANS, CGI - I, CGI - S, CDSS, GAF and QoL scale

SECONDARY OUTCOMES:
SWN, UKU, illicit substance use, laboratory measures, altered drop-out rates

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Berger, MD, Principal Investigator — ORYGEN Research Centre/ ORYGEN Youth Health
Locations (1):
- Research Sites, Melbourne, Australia

REFERENCES:
- [Derived] Hides L, Cotton SM, Berger G, Gleeson J, O'Donnell C, Proffitt T, McGorry PD, Lubman DI. The reliability and validity of the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in first-episode psychosis. Addict Behav. 2009 Oct;34(10):821-5. doi: 10.1016/j.addbeh.2009.03.001. Epub 2009 Mar 6. PMID 19324499
- [Derived] Berger GE, Proffitt TM, McConchie M, Kerr M, Markulev C, Yuen HP, O'Donnell C, Lubman D, Polari A, Wood S, Amminger PG, McGorry PD. Dosing quetiapine in drug-naive first-episode psychosis: a controlled, double-blind, randomized, single-center study investigating efficacy, tolerability, and safety of 200 mg/day vs. 400 mg/day of quetiapine fumarate in 141 patients aged 15 to 25 years. J Clin Psychiatry. 2008 Nov;69(11):1702-14. Epub 2008 Nov 18. PMID 19036233